CLINICAL TRIAL: NCT06941688
Title: Phase II, Multicentre, Randomized Study of Decitabine Plus GemOx Versus GemOx for Relapsed/Refractory Peripheral T-cell Lymphoma
Brief Title: Evaluating the Effectiveness of Decitabine With Gemcitabine, Oxaliplatin for Relapsed/Refractory Peripheral T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1904-052-1027
Record Dates: First submitted 2025-04-15; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Peripheral T-cell Lymphoma (PTCL)
Keywords: PTCL; Decitabine; GemOx; Randomized Phase II trial
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decatabine + GemOx (gemcitabine, oxaliplatin) (Experimental)
  Interventions: Drug: Decitabine with GemOx
- GemOx (gemcitabine, oxaliplatin) (Active Comparator)
  Interventions: Drug: GemOx

INTERVENTIONS:
Drug: Decitabine with GemOx — Each treatment cycle consists of 3 weeks, and a total of 6 cycles will be administered. The drugs will be administered sequentially in the following order: decitabine, gemcitabine, and oxaliplatin. Decitabine will be administered at a dose of 7.5 mg/m² on days 1 to 5; gemcitabine at 1000 mg/m² on days 1 and 8; and oxaliplatin at 100 mg/m² on day 1 of each cycle.
  Arms: Decatabine + GemOx (gemcitabine, oxaliplatin)
Drug: GemOx — Each treatment cycle spans 3 weeks, with a total of 6 cycles planned. Gemcitabine will be administered at a dose of 1000 mg/m² on days 1 and 8, and oxaliplatin at 100 mg/m² on day 1 of each cycle.
  Arms: GemOx (gemcitabine, oxaliplatin)

SUMMARY:
To establish an optimal therapeutic strategy for patients with peripheral T-cell lymphoma (PTCL) who have relapsed after first-line chemotherapy or are refractory to initial treatment, we designed a phase II trial to evaluate the efficacy of a multidrug combination regimen comprising decitabine, gemcitabine, and oxaliplatin as a second-line or later treatment. This clinical trial is based on a review of existing literature, which supports the rationale for using this three-drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be considered eligible.

  1. Patients with histologically confirmed peripheral T-cell lymphoma (PTCL) who have either relapsed after first-line chemotherapy or experienced disease progression due to refractory disease, and who are deemed eligible for further chemotherapy.
  2. Age ≥ 19 years.
  3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
  4. Adequate bone marrow function, defined as:

     1. White blood cell count ≥ 3,000/μL
     2. Absolute neutrophil count ≥ 2,000/μL
     3. Platelet count ≥ 75,000/μL
     4. Hemoglobin ≥ 8.0 g/dL Note: Transfusions within 1 week prior to screening are not permitted.
  5. Adequate renal function, defined as serum creatinine ≤ 1.5 × upper limit of normal (ULN).
  6. Adequate hepatic function, defined as:

     1. Serum total bilirubin ≤ 1.5 × ULN
     2. AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN (or ≤ 5 × ULN in the presence of liver metastases) Note: Patients with hepatic dysfunction due to underlying disease may be enrolled at the investigator's discretion.
  7. Presence of measurable disease.
  8. Ability to understand and provide written informed consent.
  9. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
  10. Female patients of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) test within 3 weeks prior to treatment, and must agree to use effective contraception (e.g., barrier methods) from 4 weeks prior to treatment initiation through the study duration.

Exclusion Criteria:

* Patients will be deemed ineligible if they meet any of the exclusion criteria listed below.

  1. Diagnosis of a malignancy other than lymphoma within the past 3 years.
  2. More than two prior lines of chemotherapy for lymphoma. Note: Autologous stem cell transplantation is considered part of one treatment regimen.
  3. Evidence of uncontrolled central nervous system involvement.
  4. History of solid organ or allogeneic stem cell transplantation.
  5. Uncontrolled seizures or significant psychiatric disorders.
  6. Pregnancy or breastfeeding.
  7. Any other serious illness or medical condition deemed inappropriate by the investigator.
  8. Presence of grade ≥2 peripheral neuropathy.
  9. Prior treatment with gemcitabine for lymphoma.
  10. History of HIV infection or active, uncontrolled bacterial, viral, or fungal infections.
  11. Surgery within 14 days prior to enrollment, or failure to recover from surgical complications.
  12. Patients currently receiving thoracic radiotherapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Objective response rate | From cycle 1 day 1 to completion of cycle 6 (each cycle is 21 days)
  The objective response rate (ORR) is defined as the proportion of patients who achieve either a complete response (CR) or a partial response (PR) to treatment, as assessed by Lugano criteria.

SECONDARY OUTCOMES:
Complete response (CR) rate | From cycle 1 day 1 to completion of cycle 6 (each cycle is 21 days)
Time to response (TTR) | From cycle 1 day 1 to completion of cycle 6 (each cycle is 21 days)
Progression-free survival (PFS) | From cycle 1 day 1 to study completion, an average of 2 years.
Overall survival (OS) | From cycle 1 day 1 to study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No